CLINICAL TRIAL: NCT02550366
Title: Novel Accelerated Contrast-Enhanced High Resolution Whole Heart Cardiac MR for Non-Invasive Evaluation of Coronary Artery Disease
Brief Title: Accelerated Contrast-Enhanced High Resolution Whole Heart Cardiac MRI
Status: Terminated | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CMR_CE_WH_AccMRI
Record Dates: First submitted 2015-08-27; First posted 2015-09-15 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Disease
Keywords: Cardiac MRI; Accelerate imaging; coronary artery disease
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CMR: Subjects with no contraindication to magnetic resonance imaging, who will undergo cardiac MRI scanning.
  Interventions: Drug: MRI Contrast

INTERVENTIONS:
Drug: MRI Contrast — MRI Contrast

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death in the United States. Cardiac MRI is a non-invasive non-ionizing technique for a comprehensive cardiac exam, which can be used in the diagnosis of CAD. In this work, the investigators will develop and validate techniques for accelerated cardiac MRI, offering better volumetric coverage of the heart, improved contrast, and superior spatial and temporal resolutions.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in the United States, even though significant efforts have been made in prevention and diagnosis. The clinical gold standard for diagnosis of CAD is catheter-based invasive x-ray angiography, performed more than a million times per year. Of these examinations, up to 35% have been found to have no significant stenosis, yet these patients had to go through the potential risks and complications of an invasive test that further exposes the patient to ionizing radiation and iodinated contrast. Thus, non-invasive diagnostic alternatives are highly desirable.

Cardiac MRI (CMR) provides a method for a comprehensive non-invasive cardiac exam, including contractile functional assessment (cine) to detect wall-motion abnormality, myocardial CMR perfusion for diagnosing perfusion defects, viability assessment using late gadolinium enhancement for evaluation of acute and chronic myocardial infarction, and coronary MRI for the identification of stenosis. CMR is advantageous in several respects, since it does not require ionizing radiation or iodinated contrast, thereby facilitating repeated or follow-up scanning. However, long data acquisition time remains as one of its main limitations. Several approaches have been studied to facilitate rapid CMR acquisition. Nonetheless, the acquisition time for high-resolution CMR remains long, and spatial and temporal resolution is traded off for acquisition time. Therefore, developments of methods to reduce the duration of data acquisition beyond what is available now are appealing. The investigators will develop novel reconstruction methodologies for high-resolution CMR that learn the anatomical structures in the images being reconstructed. The investigators will validate these techniques in a range of contrast-enhanced CMR imaging protocols, providing better volumetric coverage of the heart, efficient use of the contrast agents, and higher spatial and temporal resolution.

ELIGIBILITY:
Inclusion Criteria:

* "Healthy" subjects 18 years and older
* Cardiovascular disease patients referred from the Department of Cardiology, who do not meet any of the exclusion criteria.

Exclusion Criteria:

* Exclusion criteria include those associated with the use of MR as the imaging modality. Patients with pacemakers, implanted cardioverter-defibrillators, intracerebral clips or other implants that are not MR incompatible, atrial flutter or frequent atrial or ventricular ectopic activity, weight over 250 pounds, or significant claustrophobia will be excluded.
* Subjects should not have the following which may be hazardous to their health or interfere with MRI examinations: cardiac pacemaker; implanted cardiac defibrillator; carotid artery vascular clamp; intravascular stents, filters, or coils; aortic clip; internal pacing wires; vascular access port and/or catheter; Swan-Ganz catheter; shunt (spinal or intraventricular); aneurysm clip(s); neurostimulator; electrodes (on body, head, or brain);heart valve prosthesis; any type of prosthesis (eye, penile, etc.); artificial limb or joint replacement; bone growth/fusion stimulator; bone/joint pin, screw, nail, wire, plate; metal rods in bones; Harrington rods (spine); metal or wire mesh implants; wire sutures or surgical staples; insulin pump or infusion device; any metal fragments (i.e. metal shop); any implant held in place by a magnet; cochlear, otologic, or ear implant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population with no contraindication to magnetic resonance imaging
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Quantitative comparison of the proposed techniques with existing imaging techniques | 1 and 3 years
  vessel length and sharpness
infarct size, | 1 and 3 years
  quantitative measures
left and right ventricular volumes and masses, | 1 and 3 years
  quantitative measures
time-intensity-curve upslopes, | 1 and 3 years
  quantitative measures
high-resolution approaches with existing standard resolution imaging technique | 1 and 3 years
  quantitative measures

SECONDARY OUTCOMES:
presence of stenosis (yes/no dichotomous) | 1 and 3 years
  Qualitative comparison
presence of infarct (yes/no dichotomous), | 1 and 3 years
  Qualitative comparison
image quality (scores range from 1 [poor] to 4 [excellent]). | 1 and 3 years
  Qualitative comparison

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akcakaya, PhD, Principal Investigator — University of Minnesota
Locations (1):
- CMRR, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akcakaya M, Basha TA, Chan RH, Manning WJ, Nezafat R. Accelerated isotropic sub-millimeter whole-heart coronary MRI: compressed sensing versus parallel imaging. Magn Reson Med. 2014 Feb;71(2):815-22. doi: 10.1002/mrm.24683. PMID 23440946
- [Result] Akcakaya M, Basha TA, Pflugi S, Foppa M, Kissinger KV, Hauser TH, Nezafat R. Localized spatio-temporal constraints for accelerated CMR perfusion. Magn Reson Med. 2014 Sep;72(3):629-39. doi: 10.1002/mrm.24963. Epub 2013 Oct 7. PMID 24123058